CLINICAL TRIAL: NCT01681160
Title: Maggot Therapy in Diabetic Foot Ulcers
Brief Title: Study of Maggot Therapy in Diabetic Foot Ulcers
Acronym: MDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kerman Medical University (Other)
Responsible Party: Principal Investigator, Forough Pouryazdanpanah Kermani, university instructor, Kerman Medical University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 86/116
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: DIABETIC FOOT ULCERS
Keywords: MAGGOT THERAPY; DIABETIC FOOT; NURSING CARE; DRESSING
MeSH Terms: conditions — Diabetic Foot | interventions — Maggot Debridement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MAGGOT THERAPY & conventional therapy T (Experimental): Maggot therapy,ADMINISTERED TWO TIMES AS A NEW METHODS OF DRESSING in experimental group.conventional therapy ,administered two times in control group
  Interventions: Other: procedure:maggot therapy; Other: conventional therapy

INTERVENTIONS:
Other: procedure:maggot therapy — each times in maggot therapy continued for three days.wound assessment was done before and after any intervention
  Other Names: larval therapy
Other: conventional therapy — patients receive ordinary treatment for diabetic foot
  Other Names: mechanical debridement

SUMMARY:
This study was a Kind of clinical trial with equal randomization, that have been done from January 2009 to June 2011 in the AFZALIPOOR hospital endocrine ward in Kerman-Iran on 128 diabetic patient who had foot wounds.Replacement of conventional therapy by new methodes is one of the more important aims for health professional specially for nurses.One of this new treatment is maggot therapy.

ELIGIBILITY:
Inclusion Criteria:

* Have a chronic illness more than 7 weeks.
* The age of the patients between 40- 90 years old.
* Not having capillary disease (Blockage of artery, Rinold).
* Not user of anticoagulants and corticosteroids drugs.
* Patients without history of allergy to drugs and foods.
* Having diabetic type 2

Exclusion Criteria:

* patients who refer to critical clinical care unit
* patients who have amputation

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
change from baseline in BATES-JENSEN WOUND ASSESSMENT score at 3days and change from baseline in BATES-JENSEN WOUND ASSESSMENT score at 6 days | 2 years